CLINICAL TRIAL: NCT02554396
Title: A Single-Center, Double-Masked Evaluation of the Efficacy and Safety of PRX-100 (Aceclidine/Tropicamide) Ophthalmic Topical Formulation in the Treatment of Early to Moderate Presbyopia
Brief Title: Evaluation of the Efficacy and Safety of PRX-100 in the Treatment of Early to Moderate Presbyopia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LENZ Therapeutics, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRX100.FDAII
Record Dates: First submitted 2015-09-16; First posted 2015-09-18 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Presbyopia
Keywords: ophthalmology; vision; ocular
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- PRX-100 (Experimental): PRX-100 ophthalmic solution
  Interventions: Drug: PRX-100
- Placebo (Placebo Comparator): saline solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRX-100 — ophthalmic solution
  Arms: PRX-100
Drug: Placebo — saline ophthalmic solution
  Arms: Placebo

SUMMARY:
This is a one-day, randomized, double-masked, single-center evaluation of the efficacy and safety of PRX-100 ophthalmic solution compared to placebo in 20 subjects (randomized 4:1, PRX-100:placebo) to evaluate the safety of PRX-100 and the magnitude and duration of effects on improving near-vision acuity.

ELIGIBILITY:
Inclusion Criteria:

1. be 45-59 years of age of either sex and any race or ethnicity;
2. be able and willing to provide written informed consent and sign HIPAA form prior to any study procedure being performed;
3. be able and willing to follow all instructions and attend all study visits;
4. have a negative urine pregnancy test at Visit 1, if female of childbearing potential (those who have experienced menarche and who are not surgically sterilized [bilateral tubal ligation, hysterectomy or bilateral oophorectomy] or post-menopausal [12 months after last menses]) and must use adequate birth control throughout the study period. Adequate birth control is defined as hormonal - oral, implantable, injectable, or transdermal contraceptives; mechanical - spermicide in conjunction with a barrier such as condom or diaphragm; intrauterine device (IUD); or surgical sterilization of partner. For non-sexually active females, abstinence may be regarded as an adequate method of birth control;
5. be an early to moderate presbyope
6. be able and willing to avoid all disallowed medication(s) for the appropriate washout period and during the study without significant risk to the subject (see exclusion 15).

Exclusion Criteria:

1. have known contraindications or sensitivity to the use of any of the study medications(s) or their components;
2. have an active ocular infection (bacterial, viral or fungal), positive history of an ocular herpetic infection, preauricular lymphadenopathy, or ongoing, active ocular inflammation (e.g. moderate to severe blepharitis, allergic conjunctivitis, peripheral ulcerative keratitis, scleritis, uveitis) in either eye. Mild dry eye controlled with artificial tears and mild blepharitis controlled with lid scrubs is allowed;
3. have had surgical intervention (ocular or systemic) within 6 months prior to Visit 1, or planned surgical intervention within 30 days thereafter;
4. have had refractive surgery in the past;
5. have dry eye history defined as either current use of Restasis®, past history of insertion of punctual plugs, or daily use of artificial tears more than one drop per day;
6. have a known history of retinal detachment, diabetic retinopathy, or progressive retinal disease;
7. have an intraocular pressure that is less than 5 mmHg or greater than 22 mmHg, or be on any type of intraocular hypertension or any type of glaucoma topical treatment at Visit 1;
8. have red-green color blindness confirmed by Ishihara test during baseline procedures;
9. have an inability or refuse to discontinue contact lens wear 7 days prior to the study visit and during the study visit;
10. have used an investigational drug or device within 30 days of starting the study or be concurrently enrolled in another investigational drug or device study;
11. be a female of childbearing potential who is currently pregnant, nursing or planning a pregnancy; tests positive to a urine pregnancy test at Visit 1; or refuses to use an adequate method of contraception for the duration of the study;
12. have a condition or a situation, which in the Investigator's opinion, may put the subject at increased risk, confound study data, or interfere significantly with the subject's study participation, including but not limited to unstable: cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease;
13. use any of the following disallowed medications during the 2 weeks (14 days) prior to Visit 1 and during the study:

    * narcotic (opiate class) pain medication (e.g. codeine, oxycontin, Vicodin®, Tramadol®)
    * bladder medication (e.g. urecholine, bethanechol®)
    * antipsychotics
    * antidepressants
    * anticholinergics (e.g. atropine, belladonna, benztropine, dicyclomine, donepezil, hyoscyamine, propantheline, scopolamine, trihexphenidyl
    * dry mouth (e.g. salagen®), Evoxac®)
    * antihistamines or decongestants
    * artificial tear use of more than 1 drop per day
    * diagnostic medications required by the protocol are allowed;
14. report of recreational drug use (e.g. marijuana, methadone, heroin, cocaine).

Ages: 45 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
binocular assessment of uncorrected near visual acuity | day 1

SECONDARY OUTCOMES:
pupil diameter | day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States